CLINICAL TRIAL: NCT04708366
Title: Colon Cleansing Efficacy With 1L PEG Versus 2L PEG and 4L PEG for Colonoscopy Among Inpatients: A Randomized Controlled Trial
Brief Title: Colon Cleansing Efficacy With 1L vs. 2L vs. 4L-PEG for Colonoscopy Among Inpatients
Acronym: INTERPRET
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Lorenzo Fuccio, Professor of Gastroenterology, University of Bologna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: INTERPRET
Record Dates: First submitted 2020-12-29; First posted 2021-01-13 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Colon Disease
Keywords: colonoscopy; hospitalized patients; bowel preparation
MeSH Terms: conditions — Colonic Diseases | interventions — MoviPrep; Polyethylene Glycols

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 1L PEG (Experimental): Patients will be prepared with 1L-PEG-based bowel preparation.
  Interventions: Drug: NER1006
- 2L PEG (Active Comparator): Patients will be prepared with 2L-PEG-based bowel preparation.
  Interventions: Drug: MoviPrep
- 4L PEG (Active Comparator): Patients will be prepared with 4L-PEG-based bowel preparation.
  Interventions: Drug: Macrogol 400

INTERVENTIONS:
Drug: NER1006 — Patients will be randomly assigned (1:1:1) to receive 1L PEG (PLENVU; Norgine, Amsterdam, Netherlands), administered as a 2-day evening/morning split-dosing, or the 2L PEG + ascorbate preparation (2LPEG - MOVIPREP; Norgine), or the 4L PEG (SELG-ESSE; Alfasigma Bologna, Italy), both administered as a 2-day evening/morning split-dosing regimen.
  Other Names: IMP-1
  Arms: 1L PEG
Drug: MoviPrep — Patients will be randomly assigned (1:1:1) to receive 1L PEG (PLENVU; Norgine, Amsterdam, Netherlands), administered as a 2-day evening/morning split-dosing, or the 2L PEG + ascorbate preparation (2LPEG - MOVIPREP; Norgine), or the 4L PEG (SELG-ESSE; Alfasigma Bologna, Italy), both administered as a 2-day evening/morning split-dosing regimen.
  Other Names: IMP-2
  Arms: 2L PEG
Drug: Macrogol 400 — Patients will be randomly assigned (1:1:1) to receive 1L PEG (PLENVU; Norgine, Amsterdam, Netherlands), administered as a 2-day evening/morning split-dosing, or the 2L PEG + ascorbate preparation (2LPEG - MOVIPREP; Norgine), or the 4L PEG (SELG-ESSE; Alfasigma Bologna, Italy), both administered as a 2-day evening/morning split-dosing regimen.
  Other Names: IMP-3
  Arms: 4L PEG

SUMMARY:
An adequate level of bowel preparation before colonoscopy has an extremely relevant impact on lesion detection and procedure success. The inpatient status represents a well-known independent predictor for inadequate colon cleansing. A recent prospective, multicentre, Italian study among inpatients showed that an adequate colon cleansing was achieved in 60-70% of patients, far below the ideal threshold of 90%. Interestingly, a higher rate of adequate colon cleansing was reported for a very low-volume (1L) polyethylene glycol (PEG)-based preparation when compared to 4L and 2L PEG-based solutions. However, this finding has to be confirmed as the study was not controlled and the PEG-1L group was much smaller than the other two.

Aim of the present multicenter randomized controlled study will be to assess and compare the efficacy and safety of a novel very-low volume (1L) PEG-based preparation vs. standard-of-care low-volume (2L) and high-volume (4L) PEG-based purge, among inpatients who undergo colonoscopy.

DETAILED DESCRIPTION:
An adequate level of bowel preparation before colonoscopy has an extremely relevant impact on lesion detection and procedure success. The inpatient status represents a well-known independent predictor for inadequate colon cleansing. A recent prospective, multicentre, Italian study among inpatients showed that an adequate colon cleansing was achieved in 60-70% of patients, far below the ideal threshold of 90%. Such a low efficacy has several negative consequences: first, it leads to repetition of colonoscopy, therefore prolonging patients' in-hospital stay and increasing the risk of adverse events and costs; second, it augments the risk of missing colorectal lesions, negatively affecting patients' management and increasing costs due to the need for adjunctive diagnostic studies.

Current recommendations on bowel preparation among difficult-to-prepare patients are mostly based on expert opinions, the high-volume 4L polyethylene glycol (PEG)-based prep being considered as the gold standard, possibly with further additional solution. On the other hand, compliance to the bowel preparation has been related to an adequate colon cleansing, and it may be argued that inpatients might find it difficult to take high-volume purge. A recent Italian prospective multicentre study among inpatients showed similar rates of adequate bowel preparation between patients who underwent bowel preparation with and without additional solution. Interestingly, a higher rate of adequate colon cleansing was reported for a very low-volume (1L) polyethylene glycol (PEG)-based preparation when compared to 4L and 2L PEG-based solutions. However, this finding has to be confirmed as the study was not controlled and the PEG-1L group was much smaller than the other two.

Aim of the present randomized multicenter controlled study will be to assess and compare the efficacy and safety of a novel very-low volume (1L) PEG-based preparation vs. standard-of-care low-volume (2L) and high-volume (4L) PEG-based purge, among inpatients.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients scheduled for elective colonoscopy
* bowel preparation performed inside the hospital
* ≥18 years old

Exclusion Criteria:

* known or suspected ileus
* gastrointestinal obstruction
* gastric retention
* bowel perforation
* toxic colitis, or megacolon
* phenylketonuria
* glucose-6-phosphate dehydrogenase deficiency
* active intestinal bleeding
* emergency colonoscopy
* dementia or illness requiring nasogastric tube for bowel prep administration
* refusal to participate or inability to sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 846 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2022-03-15 (Estimated); Study Completion 2022-05-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with adequate colon cleansing | During the procedure.
  Efficacy will be assessed as the percentage of patients with adequate bowel cleansing, as rated according to the Boston Bowel Preparation Scale (BBPS). This scale gives 0-3 points to each of the three colonic segments (i.e. right colon, transverse colon, and left colon); 0 points are assigned for the worst segment cleansing, whereas at least 2 points stand for adequate segment cleansing. Adequate colon cleansing is defined when at least 2 points are reached in each colonic segment.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Fuccio, Principal Investigator — University of Bologna
Locations (1):
- Policlinico Sant'Orsola-Malpighi, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No